CLINICAL TRIAL: NCT05443230
Title: The Effect of Sarcopenia on the Efficacy and Prognosis of HCC Treated With Lenvatinib and Anti-PD-1 Treatment
Brief Title: Effect of Sarcopenia on HCC After Lenvatinib and Anti-PD-1 Treatment
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Eastern Hepatobiliary Surgery Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, Clinical Professor, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: sarcopenia and prognosis
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Liver Cancer; Sarcopenia
Keywords: liver cancer; sarcopenia; lenvatinib; immune therapy; prognosis
MeSH Terms: conditions — Liver Neoplasms; Sarcopenia | interventions — Walking Speed; Tomography, X-Ray Computed; Hand Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with sarcopenia
  Interventions: Diagnostic Test: gait speed; ct scan; grip strength and chair stand test
- patients without sarcopenia
  Interventions: Diagnostic Test: gait speed; ct scan; grip strength and chair stand test

INTERVENTIONS:
Diagnostic Test: gait speed; ct scan; grip strength and chair stand test — The chair stand test was administered, and the time required for the patient to stand five times from a sitting position without using the arms was measured. CT scan was to scan the patient's third lumbar level. For the gait speed test, the time that patients spent walking 8 meters on a flat indoor floor at usual walking speed was measured.Grip strength test:the dominant hand and the nondominant hand were measured twice intermittently (kg), and the average value of 4 values was obtained.

SUMMARY:
Sarcopenia is associated with the prognosis of HCC and cholangiocarcinoma. But there has been rare study focusing on the effect of sarcopenia on the prognosis of HCC treated with lenvatinib and anti-PD1.

DETAILED DESCRIPTION:
By tracking the short-term and long-term results of HCC patients treated with lenvatinib and anti-PD1,the difference of short-term results between patients with sarcopenia and patients without sarcopenia was analyzed, and the correlation between sarcopenia and short-term and long-term results of patients after systemic treatment was explored, so as to improve people's awareness of sarcopenia and pay attention to its prevention and treatment.All implementation details are based on the newest EWGSOP definition. The investigators consecutively admitted patients the questionnaire and evaluated the assessment of muscle strength (grip strength test and chair stand test), muscle quantity (L3 plane total skeletal muscle area) and physical performance (gait test) following the F-A-C-S approach, to confirm patients with sarcopenia accurately. And by tracking the short-term and long-term outcomes, the differences were analyzed and the relationship between sarcopenia and prognosis of systemic treatment was explored.

ELIGIBILITY:
Inclusion Criteria:

Patients with clinical diagnosis of liver cancer

* No cancer other than liver cancer has been diagnosed
* Age ≥18 years

Exclusion Criteria:

* Patients who could not complete the standard tests and questionnaires
* Patients received other therapies
* Patients who had other causes of muscle weakness (injury, fracture, stroke, etc.)
* Patients who missing CT data or CT scan did not reach the level of the third lumbar vertebra (L3)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of liver cancer admitted to the hepatobiliary surgery department and received standard tests and questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Short-term results | 3 months
  Post-treatment complications
Long-term results | 2 years
  Overall survival; Progression free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Gang Chen, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanna L, Nguo K, Furness K, Porter J, Huggins CE. Association between skeletal muscle mass and quality of life in adults with cancer: a systematic review and meta-analysis. J Cachexia Sarcopenia Muscle. 2022 Apr;13(2):839-857. doi: 10.1002/jcsm.12928. Epub 2022 Feb 13. PMID 35156342
- [Background] Arulananda S, Segelov E. Sarcopenia and cancer-related inflammation measurements in advanced gastric and junctional cancers-ready for prime time? Ann Oncol. 2022 Jul;33(7):669-671. doi: 10.1016/j.annonc.2022.04.008. Epub 2022 Apr 14. No abstract available. PMID 35430371
- [Background] Voron T, Tselikas L, Pietrasz D, Pigneur F, Laurent A, Compagnon P, Salloum C, Luciani A, Azoulay D. Sarcopenia Impacts on Short- and Long-term Results of Hepatectomy for Hepatocellular Carcinoma. Ann Surg. 2015 Jun;261(6):1173-83. doi: 10.1097/SLA.0000000000000743. PMID 24950264